CLINICAL TRIAL: NCT01801956
Title: The MILE Study: A Motivational, Individual and Locally Anchored Exercise Intervention Among 30-49 Year-olds With Low Levels of Cardiorespiratory Fitness. A Randomised Controlled Study in Primary Care.
Brief Title: The MILE Study: A Motivational, Individual and Locally Anchored Exercise Intervention in 30-49 Year Olds.
Acronym: MILE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-10-72-428-12
Record Dates: First submitted 2013-02-20; First posted 2013-03-01 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2013-10

CONDITIONS: Physical Activity
Keywords: Maximum oxygen uptake; Physical activity; Physical inactivity; Motivational interview; Cardiorespiratory fitness; Primary care; Community care
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Exercise; Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational interviewing (Active Comparator): A one hour motivational interview
  Interventions: Other: Motivational interview
- Physical activity (Experimental): Four motivational interviews, free membership of a sport club, virtual arena to upload training data from a GPS-watch
  Interventions: Behavioral: physical activity; Other: Motivational interview; Other: Virtual arena

INTERVENTIONS:
Behavioral: physical activity — free membership of a sport club
  Arms: Physical activity
Other: Motivational interview — Four motivational interviews by instructors of the local sport club
Other: Virtual arena — Uploading of training data from a GPS-watch to a virtual arena
  Arms: Physical activity

SUMMARY:
Background: Low levels of cardiorespiratory fitness are associated with high risk of non-communicable diseases and all-cause mortality. Physical activity level is the primary determinant of cardiorespiratory fitness in adults. However, knowledge on how to motivate people to engage in physical activity and maintain an active lifestyle is lacking. This study aims to investigate whether a motivational, individual, and locally anchored exercise intervention, in primary care, can improve cardiorespiratory fitness in 30 to 49 year olds with a low or very low cardiorespiratory fitness.

Design: Randomised controlled trial with 6 and 12 months follow-up. The primary outcome is cardiorespiratory fitness. Secondary outcomes include biochemical parameters (HbA1C, HDL- and LDL-cholesterol, and triglyceride), physical activity level (measured by accelerometer), self-reported physical activity, anthropometric parameters and health-related quality of life.

Methods: Cardiorespiratory fitness will be estimated via a maximal incremental exercise test and expressed as the index of maximum oxygen uptake per minute divided by body weight (ml O2/kg/min). A total of 236 participants, classified with a very low or low cardiorespiratory fitness at a local health check programme, (corresponding to ≤ 39 and ≤35 ml O2/kg/min. for 30-39 and 40-49 year-old men respectively and ≤33 and ≤31 ml O2/kg/min. for 30-39 and 40-49 year-old women respectively), will be randomised into two groups. The intervention group will receive 4 motivational interviews, six months membership to a sport club, and a global positioning watch to upload training activity to a social media. The comparison group will receive standard care: a one hour motivational interview. In addition to an Intention-to-treat analysis a per-protocol analysis will be performed. Effect of the intervention will be estimated by evaluating the differences in mean changes in cardiorespiratory fitness between the two groups.

Discussion:In new and innovative ways the focus of this study will be to improve cardiorespiratory fitness among a 30-49 year-old at-risk group using social media, GPS-technology, on-going personal support and individually tailored physical activity.

DETAILED DESCRIPTION:
Background It is well known that low levels of cardiorespiratory fitness are associated with a high risk of noncommunicable diseases and all cause mortality, and that improvements in cardiorespiratory fitness decreases this risk especially among the least fit (1-5). Although cardiorespiratory fitness has a genetic contribution, physical activity habits are the primary determinant of cardiorespiratory fitness in adults, and changes in physical activity levels result in changes in cardiorespiratory fitness (2,6). Thus the World Health Organization recommends adults aged between 18-64 to do at least 150 minutes of moderate-intensity aerobic physical activity or at least 75 minutes of vigorous-intensity aerobic physical activity weekly or an equivalent combination of moderate- and vigorous-intensity activity. In Denmark only an estimated 32 % fullfill these recommendations (7) and improving physical activity among this group of people is of great importance to public health.

In primary care several simple- and multicomponent physical activity interventions have been conducted in order to increase physical activity. However, the results of these interventions remain inconsistent. In addition, the content of the interventions is often unclearly described, particularly in relation to intensity and fidelity of the intervention delivery and reviews reveal how most of the studies use self-reported measures of physical activity (8,9). These issues warrant well-described intervention studies using objectively measures of physical activity and specifically designed for, and evaluated in primary care settings.

In Denmark, the "Check your health" programme is aimed at screening all individuals (n≈26,500) in the municipality of Randers aged between 30-49 years for cardiovascular disease during a 5-year period. Identifying people that are insufficiently active and people with a low cardiorespiratory fitness is one of the central objectives of the programme and this is done by self-reported and objective measures of physical activity and cardiorespiratory fitness.

To perform a successful intervention, strategies and techniques to motivate and guide people to adopt healthy choices need to be identified. Some of this may be accomplished by close supervision and personal instruction with healthcare professionals applying communication skills such as motivational interviewing (10,11), which has been found to be an effective approach to changing behaviour. This method specifically offers promise in improvement of cardiovascular health status (12).

Furthermore, a key issue will be to adopt modern technology and social media into the interventions (13). A Danish report supports this idea and concludes that particularly the 30-50 year olds, an age-group that does not always give high priority to regular physical activity due to lack of time and commitments such as job/further education and establishment of a family, are motivated by the social media and technology (14-16).

Finally, it is also suggested that physical activity interventions should be integrated into the structure of a broader range of community-based organisations e.g. sport clubs in order to offer a wide range of activities, and thereby individualise and anchor the physical activity locally (17).

Using the combination of motivational interviewning, social media, technology and the community organisations may build individual capability and organisational capacity for behaviour change, create new social norms, and promote policy and environmental changes that support higher levels of physical activity across the population in the long-term.

We therefore hypothesise that a locally anchored "primary care package" containing social media and technology, ongoing personal support and individually tailored flexible physical activity will improve cardiorespiratory fitness among 30-49 year-olds with a low cardiorespiratory fitness.

1. The design of a study evaluating the efficacy of a motivational, individual and locally anchored exercise intervention in primary care aiming to improve cardiorespiratory fitness among 30 to 49 year olds with low levels of cardiorespiratory fitness.
2. The actual intervention to a level of detail that allows its replication.

METHODS Study design The study is conducted as a single (researcher) blinded randomised controlled trial higly explanatory in attitude delivered under as optimal conditions as possible (18).

Sample size This study was calculated to detect a 3 ml/kg/minute (sd 6) difference between the intervention- and comparison group at the end of 6 months. The sample size calculation was based on unpuplished data from another randomised controlled health screening programme in Denmark showing a difference in cardiorespiratory fitness of 2,1 (sd 6) over a five year period and previous studies comparing 6 and 24 month intervention effects of a lifestyle physical activity program reporting differences between 3.64 (sd 3,5) and 1.34 (sd 3.37) ml/kg/minute respectively (19). With a power of 90 % using a two-sided p=0.05 test, a sample size of at least 85 in each group will be necessary. To accommodate non-independence within couples, we used robust variance estimation to obtain valid uncertainty estimates and an extra 6 participants in each group will be added to the sample size. Anticipating a drop-out of 30 %, a total of 118 participants will be included in each group.

Participants A volunteer sample of 236 participants with low or very low cardiorespiratory fitness will be recruited from the "Check your health" programme to the MILE-study.

Intervention group

The intervention will be a six month "primary care package" based on motivational, individual and locally anchored physical activity. The content is elaborated in the following:

Physical activity The participants will receive a six-month free membership for Randers Gymnastic Club, which is a nonprofit local sports club geographically situated in the middle of Randers municipality.The activities will take place in open classes with other members of the Randers Gymnastic Club and will be delivered by experienced trained instructors. The participants will decide themselves whether they will attend activities in Randers Gymnastic Club, or do moderate/vigorous/high intensity physical activity on their own or in other sport clubs.

Virtual software platform The participants will be required to upload training activities and pulse data at least once a week to the virtual software platform Endomondo.com via a global positioning system (GPS)-watch (Garmin Forerunner 210).

Motivational interviewing The intervention group will receive four motivational interviews - at baseline, after three weeks and after three and six months. The purpose of the interviews will be to support and guide the participants to the kind of physical activity that suits them and their everyday life.

The first interview will be a 90-minute long "face to face" interview in Randers Gymnastic Club including introduction to Randers Gymnastic Club, the GPS-watch and uploading of training data Endomondo.com.

The two ensuing interviews will be 15-minute telephone interviews including a status on the uploaded activities which the instructors will have access to, and finally a 30-minute face to face interview will be conducted. The motivational interviews will be delivered by trained fitness instructors from Randers Gymnastic Club, who have had a total of 8 hours training on the guiding principles underlying the motivational interview.

Comparison group Each participant in the comparison group will be invited to a one-hour motivational interview (11) about their current activity level, motivation and different options for increasing their physical activity level. The interview will be conducted by an experienced internationally certified coach at Randers Health Care Centre, and followed by a second meeting, if requested. This is the current standard care in the municipality.

Data analysis The primary analyses will be based on the intention-to-treat principle; however a per-protocol analysis will also be performed. Effect of the intervention on VO2max will be estimated by the difference of the mean changes after 6 and 12 months between the intervention group and the comparison group. Furthermore a subgroup analysis regarding gender will be performed. A Student t-test or nonparametric test will be used for normally and unevenly distributed data, respectively. Loss to follow-up analyses will be conducted via baseline characteristics from Check your health and Danish Registers. Results will be presented with 95% confidence intervals (CI) and p values. P values of <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 30-49 years old
* access to e-mail and internet
* a low or very low VO2max

Exclusion Criteria:

* health problems preventing participation
* on medication with a beta-blocker
* pregnancy
* alcoholism
* unable to communicate with the staff.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake | Change from baseline maximum oxygen uptake at 6 and 12 months.
  The outcome is measured by an indirectly standardized and validated max imalergometer bicycle test. The bicycle is cycled at 100 watt (women 70 watt). Every second minute the load is increased by 35 watt until the load causes fatigue. The highest load achieved, the time spent cycling at the highest load and the weight of the participant are put into a formula and the CRF is estimated

SECONDARY OUTCOMES:
Physical activity | Change from baseline physical activity at 6 and 12 months.
  Physical activity is measured by an accelerometer. The accelerometer is affixed with a plaster on the right anterior axillary line of the participant and worn day and night for 7 days.

OTHER OUTCOMES:
Biochemical variables | Change from baseline biochemical varibles at 12 months.
  This study will measure relevant plasma markers by means of a capillary test (HbA1c, HDL- and LDL-cholesterol, triglyceride).
Sedentary behavior | Change from baseline sedentary behavior at 6 and 12 months.
  Sedentary behavior is measured by an accelerometer. The accelerometer is affixed with a plaster on the right anterior axillary line of the participant and worn day and night for 7 days.
Anthropometric variables | Change from baseline antropometric variables at 12 months.
  BMI, waist and hip circumference
self-reported health | Change from baseline self-reported health at 12 months.
  SF-12 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine H Obling, St PhD, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University, Department of Public Health, Aarhus
  - Aarhus University, Aarhus

REFERENCES:
- [Derived] Obling KH, Overgaard K, Juul L, Maindal HT. Effects of a motivational, individual and locally anchored exercise intervention (MILE) on cardiorespiratory fitness: a community-based randomised controlled trial. BMC Public Health. 2019 Feb 28;19(1):239. doi: 10.1186/s12889-019-6556-0. PMID 30819145
- [Derived] Obling KH, Overgaard K, Juul L, Maindal HT. The MILE study: a motivational, individual and locally anchored exercise intervention among 30-49 year-olds with low levels of cardiorespiratory fitness: a randomised controlled study in primary care. BMC Public Health. 2013 Dec 23;13:1224. doi: 10.1186/1471-2458-13-1224. PMID 24365174